CLINICAL TRIAL: NCT01078857
Title: Small-fiber Neuropathy in Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chi-Chao, Chao, Department of Neurology, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200812088R
Record Dates: First submitted 2010-02-28; First posted 2010-03-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Small-Fiber Neuropathy; Chronic Kidney Disease
Keywords: Chronic kidney disease; Small-fiber neuropathy; Skin biopsy; Contact heat evoked potential; Autonomic neuropathy; Neuropathy in late stage chronic kidney disease
MeSH Terms: conditions — Small Fiber Neuropathy; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Skin biopsy — A 3-mm-diameter skin biopsy punch was taken at the lateral side of the distal leg and fixed in 4% paraformaldehyde overnight. Sections of 50 m perpendicular to the dermis were cut on a sliding microtome, quenched with 1% H2O2 in methanol, and blocked with 5% normal goat serum. Sections were incubated with rabbit antiserum to protein gene product 9.5 (PGP 9.5, UltraClone, Isle of Wight, UK, 1:1000) overnight. PGP 9.5 is a ubiquitin carboxyl hydrolase, which labels myelinated and unmyelinated nerve fibers in the peripheral nervous system. Sections were then incubated with biotinylated goat anti-rabbit immunoglobulin G (Vector, Burlingame, CA) for 1 h and the avidin-biotin complex (Vector) for another hour. The reaction product was demonstrated using chromogen SG (Vector).

SUMMARY:
Neurological dysfunction is a common complication of late stage chronic kidney disease (CKD) and peripheral nerve system is often involved in such complication. Sensory disturbances such as paresthesia and hypoesthesia are the predominant symptoms in uremic polyneuropathy and it is traditionally thought the uremic polyneuropathy mainly involve large-diameter sensory nerves. However in uremic patients the abnormal thermal thresholds, the sensory symptoms like numbness, burning, paradoxical heat, cold or freezing, and pain, and the frequent symptoms of autonomic dysfunction suggest that small-fiber neuropathy should be a clinical entity in patients of CKD. But there are still few investigations with emphasis on the changes of small-fiber nerves in CKD, and little is known about the characteristics and mechanism of small-fiber neuropathy in CKD. Skin biopsy with evaluation of epidermal nerve density and the morphology of epidermal nerves and the subepidermal nerve plexus is an effective and minimally invasive test for assessment of small-fiber neuropathy. Contact heat evoked potential (CHEP) recording the brain responses evoked by contact heat stimuli on the skin is a non-invasive technique to investigate the thermo-nociceptive pathways mediated by small-fiber nerves. In the current study, we will use an integrated approach by combining the skin biopsy, quantitative sensory testing, autonomic function tests, and CHEP to investigate the pathological, psychophysical and physiological aspects of small-fiber neuropathy in patients of CKD. The aims of the current study is to address the following issues: (1) the changes of small fiber nerves in uremia and CKD of different stage; (2) the correlation of skin innervation with clinical manifestations, thermal thresholds, and autonomic function; (3) the influence of dialysis therapy, the type of dialysis therapy, or renal transplantation on the small fiber neuropathy in uremia; (4) the roles of blood chemical substances, metals, and endocrine profiles on the development of small-fiber neuropathy; (5) the relationship between the small-fiber neuropathy and pruritus or restless leg syndrome; and (6) the pathological and physiological correlates of painful symptoms by skin biopsy and CHEP in CKD related neuropathy. The results of the study will provide important insights in the understanding of the pathogenesis, and the prevention and new treatments of small-fiber neuropathy in CKD.

ELIGIBILITY:
Inclusion Criteria:

* The patients should fulfill the criteria of CKD according to renal function study and the patients of end-stage renal disease should receive regular dialysis therapy and follow-up at outpatient clinics.
* For disease comparison, patients with peripheral neuropathy of variable etiologies will also be recruited.

Exclusion Criteria:

* Poor control DM,
* Severe heart failure,
* Bleeding tendency,
* Severe lung disease with respiratory distress,
* Severe infection,
* Alcoholism,
* Amyloidosis,
* Poor wound healing history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
The pathology of skin biopsy | within 3 months after inclusion
Intraepidermal fiber density | within 3 months after inclusion
Autonomic function | within 3 months after inclusion

SECONDARY OUTCOMES:
Function of small-fiber sensory nerve | within 3 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Tsang Hsieh, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan